CLINICAL TRIAL: NCT05251350
Title: Incarcerated Right Inguinal Hernia Containing Sigmoid Colon: An Unusual Case Report
Status: Completed | Type: Observational
Sponsor: Ahmadullah Danish (Other)
Responsible Party: Sponsor-Investigator, Ahmadullah Danish, Ahmadullah Danish, principle investigator, Kabul University of Medical Sciences
Organization: Kabul University of Medical Sciences (Other)
Other Study IDs: 2717
Record Dates: First submitted 2022-01-15; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Incarcerated Inguinal Hernia
Keywords: Incarcerated right inguinal hernia, right side, sigmoid colon
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- An incarcerated right inguinal hernia containing sigmoid colon
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — our study is observational and we use secondary data

SUMMARY:
Incarcerated inguinal hernia is an irreducible but the blood supply to the contained part is intact, but developing towards strangulation. Here the lumen of the portion of colon occupying a hernia sac is blocked with faeces.

DETAILED DESCRIPTION:
A special data collection sheet designed to collect data regarding the diagnosis, age, sex and treatment from the profile of patient retrospectively. Data entry was performed by using Microsoft Excel and all the data were analysed by SPSS.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia that requires emergency operation

Exclusion Criteria:

* hernia does not need emergency operation.

Max Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An incarcerated right inguinal hernia containing sigmoid colon.
Sampling Method: Non-Probability Sample
Enrollment: 2717 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Frequency of incarcerated right inguinal hernia containing sigmoid colon | 2013-2021
  Frequency of incarcerated right inguinal hernia containing sigmoid colon in general surgery ward of Aliabad teaching hospital, retrospectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmadullah Danish, Kabul, Afghanistan

IPD SHARING:
Plan to Share IPD: Yes